CLINICAL TRIAL: NCT05152277
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Study in Healthy Subjects to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Administered HRS9531
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HRS9531 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HRS9531-101
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: HRS9531 compared with placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single dose escalation of HRS9531 injection in healthy subjects (Experimental)
  Interventions: Drug: HRS9531
- Single dose of placebo in healthy adults (Placebo Comparator)
  Interventions: Other: placebo
- Multiple dose escalation of HRS9531 injection in healthy subjects (Experimental)
  Interventions: Drug: HRS9531
- Multiple dose of placebo in healthy adults (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: HRS9531 — Administered SC once
  Arms: Single dose escalation of HRS9531 injection in healthy subjects
Other: placebo — Administered SC once
  Arms: Single dose of placebo in healthy adults
Drug: HRS9531 — Administered SC for multiple dose
  Arms: Multiple dose escalation of HRS9531 injection in healthy subjects
Other: placebo — Administered SC for multiple dose
  Arms: Multiple dose of placebo in healthy adults

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple subcutaneous injections of HRS9531 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent;
2. Age 18-55 years on the date of signing informed consent (inclusive);
3. Body weight ≥50 kg, body mass index (BMI) within the range of 19.0-35.0 kg/m2 (inclusive);
4. Subjects with good general health, no clinically significant abnormalities.

Exclusion Criteria:

1. With previous major organ diseases, including but not limited to neuropsychiatric, cardiovascular, digestive, respiratory, urinary, endocrine, blood, immune and other diseases, are judged by researchers to be unsuitable for the study;
2. Had a severe trauma or major surgery within 6 months prior to screening, planned to undergo surgery during the trial period;
3. Participants in clinical trials of any drug or medical device in the 3 months prior to screening;
4. Blood donation history or blood loss ≥400 mL within 1 month before screening, or received blood transfusion within 2 months;
5. Allergic constitution includes severe drug allergy or history of drug allergy;
6. Hepatitis B surface antigen (HBsAg), HIV antibody detection, treponema pallidum specific antibody detection, hepatitis C virus antibody (HCVAb) positive;
7. Breast-feeding women;
8. The investigator considers that the subject has any other factors that would make it inappropriate to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Start of Treatment to end of study (approximately 7 weeks or 9 weeks)
  A summary of adverse events, including Serious Adverse Events(SAEs)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of HRS9531 | Start of Treatment to end of study (approximately 7 weeks)
  AUC of HRS9531 after single subcutaneous injection
Immunogenicity qualitative | Start of Treatment to end of study (approximately 7 weeks)
  anti-HRS9531 antibody
AUC of HRS9531 | Start of Treatment to end of study (approximately 9 weeks)
  AUC of HRS9531 after multiple subcutaneous injections
Immunogenicity qualitative | Start of Treatment to end of study (approximately 9 weeks)
  anti-HRS9531 antibody
Glucose concentration | Start of Treatment to end of study (approximately 9 weeks)
  fasting plasma glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided